CLINICAL TRIAL: NCT04448847
Title: Discovering the Mechanisms of Action for the In-vivo Protection of Aspirin-induced Enteropathy by Bifidobacterium Breve Bif195 in Man - a Randomised, Double-blinded, Placebo-controlled, Cross-over Trial in Healthy Volunteers
Brief Title: Mapping the MoA Behind GI Protection From Bif195
Acronym: PIP-M
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chr Hansen (Industry)
Responsible Party: Sponsor
Organization: ChrHansen (Unknown)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HND-GI-036
Record Dates: First submitted 2020-06-24; First posted 2020-06-26 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: Reduction of Small Intestinal Ulceration Risk

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: a randomised, double-blinded, placebo-controlled, cross-over trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo arm (Placebo Comparator): Placebo arm. Similar trial product, but without Bif195 bacteria
  Interventions: Other: Placebo
- Bif195 arm (Experimental): Active trial product with minimum 100 billion CFU daily dose
  Interventions: Dietary Supplement: Bif195

INTERVENTIONS:
Dietary Supplement: Bif195 — Active trial product with minimum 100 billion CFU daily dose
  Arms: Bif195 arm
Other: Placebo — Placebo similar to trial product but without Bif195
  Arms: Placebo arm

SUMMARY:
The trial will investigate effects of daily intake of the bacterial strain Bif195 or placebo when co-administered to once-daily oral intake of 300 mg of Acetylsalicylic Acid (ASA).

The trial includes a run-in period of two weeks duration followed by a 4-week intervention period in which Bif195/placebo and ASA are co-administered. This period is followed by a 6-week wash-out period before a new 4-week period is performed with a cross-over Bif195/placebo intervention as well as ASA co-administration. Bif195 and placebo interventions are performed double-blinded in randomised order in a cross-over fashion for each subject.

DETAILED DESCRIPTION:
Subjects will participate in the trial for a total duration of approximately 17 weeks including the run-in phase. Besides the screening visit, the trial will consist of 4 visits.

After having given their written informed consent, subjects will complete the screening procedures to evaluate their eligibility for participation in the trial and complete a run-in period of two weeks duration to washout possible pre-trial probiotics and/or use of medication. On the morning of day 4 after baseline assessments at Visit 2, all subjects will start daily intake of 300 mg ASA in combination with Bif195 or placebo in a ratio of 1:1 according to the randomisation performed at Visit 2.

At visit 2 - 5, all subjects will be biopsied from the upper small intestine and the ventricle during a gastroscopy procedure. At each of these 4 visits, 6 biopsies will be taken from pre-specified locations in the duodenum and 2 biopsies will be taken from the ventricle (approximately 5 mg each). Luminal fluids will also be collected during the gastroscopy (approximately 2 ml per visit). One venous blood sample (of 20 ml per visit) will also be collected at each of these visits.

The analysis on biopsies and luminal fluid samples will include a combination of transcriptomic, microbiome, proteomics and metabolomics analysis.

ELIGIBILITY:
Inclusion Criteria:

* • Written informed consent

  * Healthy and without any gastrointestinal discomfort/pain or other significant symptoms
  * Age ≥ 18 and ≤ 40 years
  * Willing to abstain from any other probiotic products and/or medication known to alter gastrointestinal function throughout the participation of the trial

Exclusion Criteria:

-

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2020-06-08 (Actual); Primary Completion 2021-01-12 (Actual); Study Completion 2021-01-12 (Actual)

PRIMARY OUTCOMES:
The effects of daily intake of Bif195 versus placebo | before vs after 4 week intervention
  Lanza Score obtained during endoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Filip Knop, Professor, Principal Investigator — Center for Clinical Metabolic Research, Gentofte Hospital
Locations (1):
- Center for Clinical Metabolic Research, Gentofte Hospital, Hellerup, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lon N, Engel S, Damholt A, Mortensen B, Haaber AB, Wellejus A, Knop FK. Bifidobacterium breve Bif195 ameliorates aspirin-induced gastric mucosal damage: A randomised, double blind, placebo-controlled crossover trial. Aliment Pharmacol Ther. 2024 Feb;59(3):341-349. doi: 10.1111/apt.17817. Epub 2023 Nov 30. PMID 38036761

DOCUMENTS (2):
  • Study Protocol (2020-02-18): https://cdn.clinicaltrials.gov/large-docs/47/NCT04448847/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-12): https://cdn.clinicaltrials.gov/large-docs/47/NCT04448847/SAP_001.pdf